CLINICAL TRIAL: NCT05559307
Title: Analyzing the Pharmacodynamic Substances and the Effects of Xingnaojing for Mild-to-Severe Acute Ischemic Stroke (PUBLISH): A Non-randomized, Open-label, Controlled Trial
Brief Title: Analyzing the Pharmacodynamic Substances and the Effects of Xingnaojing for Mild-to-Severe Acute Ischemic Stroke
Acronym: PUBLISH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ying Gao (Other)
Collaborators: Beijing Chaoyang Integrative Medicine Rescue and First Aid Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018YFC1705001-05-02
Record Dates: First submitted 2021-11-11; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke | interventions — xingnaojing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xingnaojing injection group (Experimental): Subjects will receive intravenously administered Xingnaojing injection, combined with guidelines-based standard care.
  Interventions:
  Drugs:Xingnaojing injection Other: Standard care (eg. antiplatelet drugs and statins)
  Interventions: Drug: Xingnaojing injection
- Standard care group (No Intervention): Subjects will receive guidelines-based standard care.
  Interventions:
  Other: Standard care (eg. antiplatelet drugs and statins)

INTERVENTIONS:
Drug: Xingnaojing injection — Xingnaojing injection 20 ml+0.9% diluted sodium chloride injection 250ml, IV (in the vein), every 12 hours for 7 days.
  Arms: Xingnaojing injection group

SUMMARY:
The main purposes of this trial are to analyze the pharmacodynamic substances and the effects of Xingnaojing for mild-to-severe acute ischemic stroke.

DETAILED DESCRIPTION:
Xingnaojing is widely used in China, but there is lack of sufficient and reasonable explanation of its intervention effects for acute ischemic stroke currently. In order to further clarify the main pharmacodynamic substances of Xingnaojing in the treatment of acute ischemic stroke, this study intends to carry out a non-randomized, open-label, controlled clinical trial. The primary hypothesis is that , compared with the control group, Xingnaojing will produce serial changes in plasma metabolites at baseline (pre-dose) and 7 days, as well as urine metabolites at baseline (pre-dose), 6 days, 7 days and 8 days. The serial changes may be the potential support to explain the intervention effect of Xingnaojing. All participants will have a National Institutes of Health Stroke Scale(NIHSS)entry score of 4-25. Participants who have planned or already received the intravenous thrombolysis or endovascular treatment will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute ischemic stroke；
* Symptom onset within 24 hours；
* 40 ≤ age ≤ 80 years;
* 4 ≤ NIHSS ≤ 25；
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Planned or already receiving intravenous thrombolysis or endovascular treatment;
* Suspected secondary stroke caused by tumor, brain trauma, or hematological diseases;
* Already dependent in activities of daily living before the present acute stroke (defined as modified Rankin Scale score ≥ 2) ;
* Other conditions that cause cardiogenic embolism (e.g., atrial fibrillation, rheumatic heart disease, valvular heart disease);
* Other conditions that lead to motor dysfunction (e.g., severe osteoarthrosis, rheumatoid arthritis);
* Significant renal or hepatic insufficiency (defined as a serum creatinine concentration, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) value that is twice the upper limit of normal);
* Life expectancy of 3 months or less due to other life-threatening illness (e.g.,advanced cancer)
* Other conditions that render outcomes or follow-up unlikely to be assessed;
* Known to be pregnant or breastfeeding;
* Use any drugs containing traditional Chinese medicine within 1 week before enrollment;
* Currently receiving an investigational drug.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Differences in Borneol, Muscone, 1,8-Cineole between Xingnaojing injection group and standard care group at baseline. | Baseline
  Differences in the content of Borneol, Muscone, 1,8-Cineole in plasma and urine samples between Xingnaojing injection group and standard care group at baseline.
Differences in Borneol, Muscone, 1,8-Cineole between Xingnaojing injection group and standard care group at 6 days. | 6 days
  Differences in the content of Borneol, Muscone, 1,8-Cineole in plasma and urine samples between Xingnaojing injection group and standard care group at 6 days.
Differences in Borneol, Muscone, 1,8-Cineole between Xingnaojing injection group and standard care group at 7 days. | 7 days
  Differences in the content of Borneol, Muscone, 1,8-Cineole in plasma and urine samples between Xingnaojing injection group and standard care group at 7 days.
Differences in Borneol, Muscone, 1,8-Cineole between Xingnaojing injection group and standard care group at 8 days. | 8 days
  Differences in the content of Borneol, Muscone, 1,8-Cineole in plasma and urine samples between Xingnaojing injection group and standard care group at 8 days.

SECONDARY OUTCOMES:
The change of neurological deficits | Baseline, 7 days
  The change of neurological deficits is measured by the change of National Institute of Health Stroke Scale (NIHSS) score, ranging from 0 (best score) to 42 (worst score).
Patient reported outcome | 7 days
  Patient reported outcome is measured by Patient reported outcome (PRO) scale of stroke, ranging from 0(worst score) to 180 (best score).
The proportion of life dependency | 30 days, 90 days
  The proportion of life dependency is defined as Modified Rankin Scale (mRS) score 0-2. The mRS score ranges from 0 (best score) to 6 (worst score).
The degree of disability | 30 days, 90 days
  The degree of disability is measured by the distribution proportion of mRS score, ranging from 0 (best score) to 6 (worst score).
Number of participants with cerebral vascular incidents | 90 days
  Cerebral vascular incidents are defined as stroke, transient ischemia attack, etc.
Number of participants with cardio-cerebral vascular incidents | 90 days
  Cardio-cerebral vascular incidents are defined as stroke, acute coronary syndrome (acute ST-elevation myocardial infarction, acute non-ST-elevation myocardial infarction and unstable angina), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Gao, Principal Investigator — Dongzhimen Hospital
Locations (1):
- Beijing Chaoyang Integrative Medicine Rescue and First Aid Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No